CLINICAL TRIAL: NCT02536183
Title: A Phase I Study of Lyso-thermosensitive Liposomal Doxorubicin (LTLD, ThermoDox®) and Magnetic Resonance-Guided High Intensity Focused Ultrasound (MR-HIFU) for Relapsed or Refractory Solid Tumors in Children, Adolescents, and Young Adults
Brief Title: A Phase I Study of Lyso-thermosensitive Liposomal Doxorubicin and MR-HIFU for Pediatric Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: AeRang Kim (Other)
Responsible Party: Sponsor-Investigator, AeRang Kim, MD, PhD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU Thermodox
Record Dates: First submitted 2015-08-13; First posted 2015-08-31 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Pediatric Cancer; Solid Tumors; Rhabdomyosarcoma; Ewing Sarcoma; Soft Tissue Sarcomas; Osteosarcoma; Neuroblastoma; Wilms Tumor; Hepatic Tumor; Germ Cell Tumors
Keywords: Solid tumors; relapsed pediatric solid tumors; high intensity focused ultrasound; Lyso-thermosensitive liposomal doxorubicin; ThermoDox; relapsed sarcoma; Ewing Sarcoma family of tumors; Osteosarcoma; Neuroblastoma; Wilms Tumor; Hepatic Tumor; Germ Cell Tumors
MeSH Terms: conditions — Neoplasms; Rhabdomyosarcoma; Sarcoma, Ewing; Sarcoma; Osteosarcoma; Neuroblastoma; Wilms Tumor; Carcinoma, Hepatocellular; Neoplasms, Germ Cell and Embryonal; Neuroectodermal Tumors, Primitive, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): LTLD will be administered intravenously in combination with MR-HIFU ablation on day 1 of every 21 day cycle. There will be two potential dose escalation of LTLD with highest dose not to exceed the adult recommended MTD. Patients may receive up to a total of 6 cycles.
  Interventions: Device: Magnetic resonance high intensity focused ultrasound; Drug: Lyso-thermosensitive liposomal doxorubicin
- Part B (Experimental): LTLD at dose determined from Part A will be administered intravenously on day 1 of every 21 day cycle. MR-HIFU induced MHT will follow immediately post LTLD infusion for one hour to target area with target temperatures of 40-45°C. Patients may receive up to a total of 6 cycles
  Interventions: Device: Magnetic resonance high intensity focused ultrasound; Drug: Lyso-thermosensitive liposomal doxorubicin

INTERVENTIONS:
Device: Magnetic resonance high intensity focused ultrasound — Magnetic resonance (MR)-high intensity focused ultrasound (HIFU) provides precise controlled delivery of heat by focusing ultrasound energy inside a lesion using an external applicator that is completely non-invasive and non-ionizing.
  Other Names: MR-HIFU
Drug: Lyso-thermosensitive liposomal doxorubicin — A heat-activated formulation of liposomal doxorubicin with unique property of heat-activated release of doxorubicin, an active agent in most pediatric solid tumors.
  Other Names: LTLD; ThermoDox

SUMMARY:
This study is looking to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of lyso-thermosensitive liposomal doxorubicin (LTLD) administered in combination with MR-HIFU in children with relapsed/refractory solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing's sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms' tumor, hepatic tumors, and germ cell tumors.

DETAILED DESCRIPTION:
This is phase 1 trial of LTLD with MR-HIFU induced heating in children and young adults with relapsed/refractory solid tumors.

Part A of the trial will be a traditional dose escalation study to determine the pediatric MTD/RP2D of LTLD combined with MR-HIFU ablation which allows for release of doxorubicin in the ablation zone and peri-ablation margins.

Part B of the trial will combine LTLD at the MTD/RP2D with MR-HIFU induced mild hyperthermia (MHT) in an expanded cohort.

ELIGIBILITY:
Inclusion Criteria:

Part A: ≤21 years of age Part B: ≤ 30 years of age.

DIAGNOSIS:

Histologically confirmed malignant solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing's sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms' tumor, hepatic tumors, germ cell tumors.

TUMOR LOCATION:

Patient must have at least one tumor located in areas accessible to HIFU, which will be defined as the target lesion(s). Target lesions must be reachable within the normal safety margins of HIFU as specified in the instructions for use.

TARGET LESION(S):

Radiographically evaluable or measurable solid tumor target lesion(s).

THERAPEUTIC OPTIONS:

Malignant Tumor: The patient's cancer must have relapsed after or failed to respond to frontline curative therapy and there must not be other potentially curative treatment options available.

PRIOR THERAPY:

Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering on this study.

No limitation on the number of prior chemotherapy regimens that the patient may have received prior to study entry.

Myelosuppressive chemotherapy: The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks prior to study entry. Prior treatment with anthracyclines is allowed as long as total cumulative dose is ≤ 450 mg/m2.

Immunotherapy: The last dose of immunotherapy (monoclonal antibody or vaccine) must be at least 4 weeks prior to study entry.

Biologic (anti-cancer agent): The last dose of all biologic agents for the treatment of the patient's cancer (such as retinoids or tyrosine kinase inhibitors) must be at least 7 days prior to study entry.

Radiation therapy: The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry. The last dose of all other local palliative (limited port) radiation must be at least 2 weeks prior to study entry.

Stem Cell Transplantation. At least 2 months post-autologous stem cell transplant or at least 3 months post-allogeneic transplant and recovered from toxicities without evidence of graft versus host disease and on stable doses of immunosuppressive medications if required.

Growth Factors. The last dose of colony stimulating factors, such as filgrastim, sargramostim, and erythropoietin, must be at least 1 week prior to study entry. The last dose of long-acting colony stimulating factors, such as peg-filgrastim, must be at least 2 weeks prior to study entry.

CONCURRENT THERAPIES:

No other anti-cancer therapy (chemotherapy, biological therapy, radiation therapy) is permitted.

PERFORMANCE STATUS:

Patients > 16 years old must have a Karnofsky performance level ≥ 50%, and children ≤ 16 years old must have a Lansky performance level ≥ 50%.

HEMATOLOGIC FUNCTION:

Peripheral absolute neutrophil count (ANC) of ≥1000/µL. Platelet count ≥75,000/µL (transfusion independent (no transfusion within at least 7 days prior to enrollment)).

HEPATIC FUNCTION:

Total bilirubin must be ≤ 1.5 times the upper limit of normal (ULN) for age and gender. SGPT (ALT) must be ≤ 3.0 times the upper limit of normal for age.

RENAL FUNCTION:

Age-adjusted normal serum creatinine OR a creatinine clearance ≥ 60 mL/min/1.73 m2.

CARDIAC FUNCTION:

Adequate Cardiac Function with Ejection Fraction > 50% by echocardiogram or cardiac MRI within 14 days prior to starting therapy.

Exclusion Criteria:

Clinically significant unrelated systemic illness, such as serious infections, hepatic, renal or other organ dysfunction, which in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate study interventions.

Patients who are pregnant or breast-feeding are not eligible for this study due to risks of fetal and teratogenic adverse events seen in animal/human studies with doxorubicin. Negative pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive methods beginning at the signing of informed consent and until at least 30 days after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or designated associate.

Implant or prosthesis or scar tissue within the path of the HIFU beam.

Target lesion <1 cm from nerve plexus, spinal canal, and bowel.

Target lesion in contact with hollow viscera.

Lesion in the skull.

Inability to undergo MRI and/or contraindication for MRI.

Inability to tolerate stationary position during HIFU.

Previous history of hypersensitivity to doxorubicin or its liposomal formulations.

Patients currently receiving other anticancer agents.

Patients currently receiving other investigational agents.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2016-10; Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of LTLD | 3 weeks
  To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of LTLD administered in combination with MR-HIFU ablation in children with relapsed/refractory solid tumors by examining blood samples collected from participants
Toxicity profile of LTLD | up to 18 weeks
  To define and describe the toxicities of LTLD administered in combination with MR-HIFU as measured by reportable adverse events of participants as per the CTCAE v 4.0
Pharmacokinetics of LTLD | 8 days
  Analyze blood samples of participants to characterize the pharmacokinetic properties of LTLD administered in combination with MR-HIFU
Feasibility of treatment | up to 18 weeks
  To determine the feasibility of LTLD administered at the recommended dose in combination with MR-HIFU induced mild hyperthermia (MHT) as determined by patient outcomes and adverse events

SECONDARY OUTCOMES:
Antitumor Activity of the Treatment | up to 18 weeks
  To preliminarily determine the antitumor activity of LTLD with MR-HIFU within the confines of a phase 1 study by examining the response of target lesions using RECIST criteria v1.1
Social Impact of the Treatment on Participants | up to 18 weeks
  To determine changes in symptoms and quality of life in children treated with LTLD and MR-HIFU by administering the Symptom Distress Scale and Peds QL v4.0 to participants
Determine the Changes in Pharmacodynamic Immune Markers in Participants | 3 weeks
  To determine the changes in immune markers in children treated with LTLD and MR-HIFU by examining blood samples from participants

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903